CLINICAL TRIAL: NCT02814643
Title: A Multicenter, Randomized, Double-blind, Parallel Group, Placebo-controlled, Phase 3b Study to Evaluate the Potential Effect of Benralizumab on the Humoral Immune Response to the Seasonal Influenza Vaccination in Adolescent and Young Adult Patients With Severe Asthma.
Brief Title: Study to Evaluate the Potential Effect of Benralizumab on the Humoral Immune Response to the Seasonal Influenza Vaccination in Adolescent and Young Adult Patients With Severe Asthma
Acronym: ALIZE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: D3250C00033
Record Dates: First submitted 2016-06-15; First posted 2016-06-28 (Estimated); Results first posted 2018-03-01 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Asthma
Keywords: Male and female adolescent patients; severe asthma
MeSH Terms: conditions — Asthma | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Benralizumab (Experimental): 1 mL fill volume administered every 4 weeks for 3 doses (Weeks 0, 4, and 8). Patients will receive 1 dose of seasonal influenza virus vaccine Intramuscular (IM) at Week 8.
  Interventions: Drug: Benralizumab; Drug: Seasonal influenza virus vaccine
- Placebo (Placebo Comparator): 1 mL fill volume administered every 4 weeks for 3 doses (Weeks 0, 4, and 8). Patients will receive 1 dose of seasonal influenza virus vaccine Intramuscular (IM) at Week 8.
  Interventions: Drug: Benralizumab Placebo; Drug: Seasonal influenza virus vaccine

INTERVENTIONS:
Drug: Benralizumab — Benralizumab SC administered every 4 weeks for 3 doses (Weeks 0, 4, and 8).
  Arms: Benralizumab
Drug: Benralizumab Placebo — Placebo administered every 4 weeks for 3 doses (Weeks 0, 4, and 8).
  Arms: Placebo
Drug: Seasonal influenza virus vaccine — Patients will receive 1 dose of seasonal influenza virus vaccine Intramuscular (IM) at Week 8.

SUMMARY:
This is a randomized, double-blind, parallel group, placebo-controlled study designed to investigate the potential effect of a fixed dose of benralizumab administered subcutaneously (SC) on antibody responses following seasonal influenza virus vaccination

DETAILED DESCRIPTION:
This study is designed to investigate the potential effect of benralizumab on the antibody response to the seasonal influenza virus vaccine in patients 12-21 years of age with asthma. Benralizumab will be given subcutaneously (SC) at Weeks 0, 4, and 8 weeks, at which time benralizumab levels will reach steady state. Patients will then receive 1 dose of intramuscular (IM) seasonal influenza virus vaccine at Week 8 and samples drawn at Week 8 and Week 12 to measure the antibody response to the influenza virus

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients aged 12 to 21 years, inclusive, at the time of Visit 1
* Weight of ≥40 kg
* Documented history of current treatment with Inhaled corticosteroids (ICS) and long-acting β2 agonists (LABA)
* Morning pre-bronchodilator forced expiratory volume in 1 second (FEV1) of >50% predicted at Visit 1 or Visit 2.
* Airway reversibility (FEV1 >12% and 200 ml) demonstrated at Visit 1 or Visit 2 using the Maximum Post-bronchodilator Procedure OR
* Airway reversibility documented in the previous 12 months prior to Visit 1
* An exacerbation, 1 or more, that required oral corticosteroids in the previous year OR
* Any condition assessed by patient recall over the previous 2-4 weeks

Exclusion Criteria:

* Clinically important pulmonary disease other than asthma
* Known history of allergy or reaction to the Investigational Product formulation or influenza vaccine
* Receipt of an influenza vaccine within 90 days prior to randomization
* Poorly controlled asthma during the screening period that requires treatment with oral corticosteroids or a hospitalization/emergency room visit for the treatment of asthma
* Acute illness or evidence of significant active infection or known influenza infection during the current flu season

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 103 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-01-24 (Actual); Study Completion 2017-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela L Zeitlin, M.D. Ph.D., Principal Investigator — Johns Hopkins University
Locations (22):
- United States (22):
  - Research Site, Birmingham, Alabama
  - Research Site, Mesa, Arizona
  - Research Site, Huntington Beach, California
  - Research Site, Newport Beach, California
  - Research Site, Aurora, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Aventura, Florida
  - Research Site, Miami, Florida
  - Research Site, Minneapolis, Minnesota
  - Research Site, Bellevue, Nebraska
  - Research Site, Northfield, New Jersey
  - Research Site, Edmond, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, North Charleston, South Carolina
  - Research Site, Arlington, Texas
  - Research Site, El Paso, Texas
  - Research Site, New Braunfels, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Waco, Texas
  - Research Site, Clinton, Utah

REFERENCES:
- See also: CSP redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3366&filename=d3250c00033-clinical-study-protocol_Redacted.pdf
- See also: Statistical Analysis Plan (SAP) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3366&filename=d3250C00033-sap-edition-2_redacted.pdf
- See also: ALIZE_redacted_protocol.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3366&filename=ALIZE_redacted_protocol.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 30 study centers in the United States between 01 July 2016 and 24 January 2017
Pre-assignment Details: The study duration was up to 23 weeks, consisting of an initial screening period lasting up to 3 weeks, a 12-week treatment period, and a follow-up visit 8 weeks after the last dose of study drug
Groups:
- Benralizumab 30mg: Benralizumab 30mg/day subcutaneous
- Placebo: Placebo to benralizumab subcutaneous
Period: Overall Study
Arm/Group | Benralizumab 30mg | Placebo
Started | 51 | 52
Completed | 50 | 49
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Benralizumab 30mg | Placebo | Total
Number analyzed (Participants) | 51 | 52 | 103
Age, Continuous [Mean (Standard Deviation); unit: Years] | 16.0 (2.65) [12 to 21] | 15.7 (2.99) [12 to 21] | 15.9 (2.82) [12 to 21]
Age, Customized [Number; unit: Participants]
  ≥12 to ≤17 | 36 | 36 | 72
  ≥18 to ≤21 | 15 | 16 | 31
Sex/Gender, Customized [Number; unit: Participants]
  Female | 21 | 21 | 42
  Male | 30 | 31 | 61
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian Or Alaska Native | 0 | 1 | 1
  Black Or African American | 13 | 13 | 26
  Other | 0 | 2 | 2
  White | 38 | 36 | 74

OUTCOME MEASURES:

1. Primary Outcome: Postdose Strain-specific Hemagglutination-inhibition (HAI) Antibody Geometric Mean Fold Rise From Week 8 to Week 12
Description: To compare the geometric mean fold rises in influenza strain-specific hemagglutination-inhibition responses from Week 8 to Week 12 between patients receiving benralizumab 30mg and patients receiving placebo. Geometric mean fold rise was defined as antilog(z) (mean [log(z) x]), where "x" is the postdose HAI antibody titer fold rise from Week 8 and "z" is the natural logarithm.
Time Frame: 4 weeks
Population: The vaccine immunogenicity analysis set included all randomized patients who received ≥1 dose of planned study drugs, had pre- (Week 8) and postdose (Week 12) HAI or microneutralization antibody measurements, and had no protocol deviations judged to have the potential to interfere with the generation or interpretation of an antibody response.
Measure: Geometric Least Squares Mean (Standard Error); unit: Fold change
Arm/Group | Benralizumab 30mg | Placebo
Number analyzed (Participants) | 50 | 49
Fold change
  Influenza A H1N1 | 3.60 (1.22) | 3.13 (1.22)
  Influenza A H3N2 | 3.25 (1.18) | 3.85 (1.18)
  Influenza B Yamagata lineage | 3.42 (1.16) | 3.17 (1.16)
  Influenza B Victoria lineage | 4.08 (1.19) | 3.27 (1.19)
Statistical Analysis 1: Comparison: Benralizumab 30mg vs Placebo; Influenza A H1N1; Test type: Other; ANCOVA; The linear model effects are treatment group as a fixed effect and age group (adolescents and young adults) as fixed categorical covariate; Geometric least-square mean ratio = 0.87, 90% CI 2-sided [0.56 to 1.35]
Statistical Analysis 2: Comparison: Benralizumab 30mg vs Placebo; Influenza A H3N2; Test type: Other; ANCOVA; [statistical method as in outcome 1, analysis 1]; Geometric least-square mean ratio = 1.19, 90% CI 2-sided [0.82 to 1.71]
Statistical Analysis 3: Comparison: Benralizumab 30mg vs Placebo; Influenza B Yamagata lineage; Test type: Other; ANCOVA; [statistical method as in outcome 1, analysis 1]; Geometric least-square mean ratio = 0.93, 90% CI 2-sided [0.67 to 1.29]
Statistical Analysis 4: Comparison: Benralizumab 30mg vs Placebo; Influenza B Victoria lineage; Test type: Other; ANCOVA; [statistical method as in outcome 1, analysis 1]; Geometric least-square mean ratio = 0.80, 90% CI 2-sided [0.54 to 1.19]

2. Primary Outcome: Postdose Strain-specific Hemagglutination-inhibition Antibody Geometric Mean Titers Obtained at Week 12
Description: To compare the geometric mean titers of hemagglutination-inhibition antibody as a measure of influenza strain-specific response at Week 12 between patients receiving benralizumab 30mg and patients receiving placebo.
Time Frame: 12 weeks
Population: The vaccine immunogenicity analysis set included all randomized patients who received at least 1 dose of planned study drugs, had pre- (Week 8) and postdose (Week 12) HAI or MN antibody measurements, and had no protocol deviations judged to have the potential to interfere with the generation or interpretation of an antibody response.
Measure: Geometric Least Squares Mean (Standard Error); unit: Antibody titer
Arm/Group | Benralizumab 30mg | Placebo
Number analyzed (Participants) | 50 | 49
Antibody titer
  Influenza A H1N1 | 521.06 (1.13) | 518.60 (1.13)
  Influenza A H3N2 | 170.73 (1.15) | 219.35 (1.15)
  Influenza B Yamagata lineage | 61.47 (1.13) | 63.15 (1.13)
  Influenza B Victoria lineage | 53.10 (1.14) | 66.85 (1.14)
Statistical Analysis 1: Comparison: Benralizumab 30mg vs Placebo; Influenza A H1N1; Test type: Other; ANCOVA; [statistical method as in outcome 1, analysis 1]; Geometric least-square mean ratio = 1.00, 90% CI 2-sided [0.76 to 1.31]
Statistical Analysis 2: Comparison: Benralizumab 30mg vs Placebo; Influenza A H3N2; Test type: Other; ANCOVA; [statistical method as in outcome 1, analysis 1]; Geometric least-square mean ratio = 1.28, 90% CI 2-sided [0.93 to 1.77]
Statistical Analysis 3: Comparison: Benralizumab 30mg vs Placebo; Influenza B Yamagata lineage; Test type: Other; ANCOVA; [statistical method as in outcome 1, analysis 1]; Geometric least-square mean ratio = 1.03, 90% CI [0.79 to 1.34]
Statistical Analysis 4: Comparison: Benralizumab 30mg vs Placebo; Influenza B Victoria lineage; Test type: Other; ANCOVA; [statistical method as in outcome 1, analysis 1]; Geometric least-square mean ratio = 1.26, 90% CI [0.93 to 1.70]

3. Primary Outcome: Proportion of Patients Who Experienced a Strain-specific Postdose Antibody Response at Week 12 With Antibody Response Defined as a ≥4-fold Rise in Hemagglutination-inhibition Antibody Titer From Week 8 to Week 12
Description: To compare the proportions of patients experiencing influenza strain-specific responses as measured by ≥4-fold rises in hemagglutination-inhibition antibody titer from Week 8 to Week 12 between patients receiving benralizumab 30mg and patients receiving placebo.
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Proportion of Participants
Arm/Group | Benralizumab 30mg | Placebo
Number analyzed (Participants) | 50 | 49
Proportion of Participants
  Influenza A H1N1 | 0.440 [0.32 to 0.57] | 0.306 [0.20 to 0.43]
  Influenza A H3N2 | 0.500 [0.38 to 0.62] | 0.490 [0.37 to 0.62]
  Influenza B Yamagata lineage | 0.480 [0.36 to 0.60] | 0.490 [0.37 to 0.62]
  Influenza B Victoria lineage | 0.560 [0.43 to 0.68] | 0.408 [0.29 to 0.54]

4. Primary Outcome: Proportion of Patients Who Achieved a Strain-specific Postdose Hemagglutination-inhibition Antibody Titer ≥40 at Week 12
Description: To compare the proportions of patients experiencing influenza strain-specific responses as measured by ≥40-fold rises in hemagglutination-inhibition antibody titer at Week 12 between patients receiving benralizumab 30mg and patients receiving placebo.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Proportion of Participants
Arm/Group | Benralizumab 30mg | Placebo
Number analyzed (Participants) | 50 | 49
Proportion of Participants
  Influenza A H1N1 | 1.00 (251.9) [0.94 to 1.00] | 1.00 (191.3) [0.94 to 1.00]
  Influenza A H3N2 | 0.980 (136.2) [0.91 to 1.00] | 0.980 (168.6) [0.91 to 1.00]
  Influenza B Yamagata lineage | 0.860 (144.9) [0.75 to 0.93] | 0.796 (115.0) [0.68 to 0.88]
  Influenza B Victoria lineage | 0.780 (178.7) [0.66 to 0.87] | 0.878 (162.2) [0.77 to 0.95]

5. Secondary Outcome: Proportion of Patients Who Achieved a Strain-specific Postdose Hemagglutination Inhibition Antibody Titre ≥320 at Week 12
Description: To compare the proportions of patients experiencing influenza strain-specific responses as measured by ≥320-fold rises in hemagglutination-inhibition antibody titer at Week 12 between patients receiving benralizumab 30mg and patients receiving placebo.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Proportion of Participants
Arm/Group | Benralizumab 30mg | Placebo
Number analyzed (Participants) | 50 | 49
Proportion of Participants
  Influenza A H1N1 | 0.840 [0.73 to 0.92] | 0.857 [0.75 to 0.93]
  Influenza A H3N2 | 0.500 [0.38 to 0.62] | 0.612 [0.48 to 0.73]
  Influenza B Yamagata lineage | 0.020 [0.00 to 0.09] | 0.020 [0.00 to 0.09]
  Influenza B Victoria lineage | 0.080 [0.03 to 0.17] | 0.041 [0.01 to 0.12]

6. Secondary Outcome: Postdose Strain-specific Microneutralization Antibody Geometric Mean Fold Rise From Week 8 to Week 12
Description: To compare the geometric mean fold rises in influenza strain-specific microneutralization antibody responses from Week 8 to Week 12 between patients receiving benralizumab 30mg and patients receiving placebo. Geometric mean fold rise was defined as antilog(z) (mean [log(z) x]), where "x" is the postdose microneutralization antibody titer fold rise from Week 8 and "z" is the natural logarithm.
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fold change
Arm/Group | Benralizumab 30mg | Placebo
Number analyzed (Participants) | 50 | 49
Fold change
  Influenza A H1N1 | 5.1 (521.4) | 4.4 (329.4)
  Influenza A H3N2 | 3.2 (149.8) | 3.6 (210.0)
  Influenza B Yamagata lineage | 2.8 (148.9) | 3.2 (141.3)
  Influenza B Victoria lineage | 3.8 (224.1) | 3.5 (195.3)

7. Secondary Outcome: Postdose Strain-specific Serum Microneutralization Antibody Geometric Mean Titers Obtained at Week 12
Description: To compare the geometric mean titers of microneutralization antibody as a measure of influenza strain-specific response at Week 12 between patients receiving benralizumab 30mg and patients receiving placebo.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Antibody titer
Arm/Group | Benralizumab 30mg | Placebo
Number analyzed (Participants) | 50 | 49
Antibody titer
  Influenza A H1N1 | 3774.1 (181.7) | 3969.1 (154.0)
  Influenza A H3N2 | 4307.5 (169.0) | 4351.3 (171.0)
  Influenza B Yamagata lineage | 350.2 (103.6) | 336.2 (114.3)
  Influenza B Victoria lineage | 164.5 (178.5) | 234.4 (135.0)

8. Secondary Outcome: Proportion of Patients Who Experience a Strain-specific Postdose Antibody Response at Week 12 With Antibody Response Defined as a ≥4-fold Rise in Microneutralization Antibody Titer From Week 8 to Week 12
Description: To compare the proportions of patients experiencing influenza strain-specific responses as measured by ≥4-fold rises in microneutralization antibody titer from Week 8 to Week 12 between patients receiving benralizumab 30mg and patients receiving placebo.
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Proportion of Participants
Arm/Group | Benralizumab 30mg | Placebo
Number analyzed (Participants) | 50 | 49
Proportion of Participants
  Influenza A H1N1 | 0.420 (251.9) [0.30 to 0.55] | 0.408 (191.3) [0.29 to 0.54]
  Influenza A H3N2 | 0.440 (136.2) [0.32 to 0.57] | 0.429 (168.6) [0.31 to 0.56]
  Influenza B Yamagata lineage | 0.280 (144.9) [0.18 to 0.40] | 0.388 (115.0) [0.27 to 0.52]
  Influenza B Victoria lineage | 0.400 (178.7) [0.28 to 0.53] | 0.388 (162.2) [0.27 to 0.52]

9. Secondary Outcome: Change From Baseline in Mean Asthma Control Questionnaire 6 (ACQ-6) Score at Week 12
Description: To compare the change from baseline at Week 12 in mean ACQ-6 score between patients receiving benralizumab 30mg and patients receiving placebo. The ACQ-6 assesses asthma symptoms (nighttime waking, symptoms on waking, activity limitation, shortness of breath, wheezing, and short-acting β2 agonist use). Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ-6 score is the mean of the responses to each question. Mean scores of ≤0.75 indicate well-controlled asthma, scores between 0.75 and ≤1.5 indicate partly controlled asthma, and a score >1.5 indicates not well controlled asthma
Time Frame: 12 weeks
Population: The full analysis set included all patients who were randomized and received any investigational product.
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Benralizumab 30mg | Placebo
Number analyzed (Participants) | 50 | 49
Score on a scale | -0.50 [-2.8 to 4.3] | -0.42 [-2.7 to 1.2]

ADVERSE EVENTS:
Time Frame: All AEs, including SAEs, were collected from the time the patient, parent, or legal guardian signed the informed consent/assent throughout the treatment period and including the follow-up period (through Week 20).
Arm/Group | Benralizumab 30mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/51 | 2/52
Other Adverse Events (participants affected / at risk) | 28/51 | 23/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benralizumab 30mg (N=51) | Placebo (N=52)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benralizumab 30mg (N=51) | Placebo (N=52)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 4 (5)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 4 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least 30 days prior to submission for publication/presentation, Institution and PI shall jointly provide AZ with material for review. No publication/presentation may include any of AZ's Confidential Information without AZ's written approval. AZ can request Institution and PI to withhold material from submission for publication/presentation for an additional 90 days to allow AZ to establish and preserve its proprietary rights in the material being submitted for publication/presentation.

DOCUMENTS (2):
  • Study Protocol (2015-12-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT02814643/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/43/NCT02814643/SAP_001.pdf